CLINICAL TRIAL: NCT05250596
Title: On-admission Low-dose Colchicine in Addition to Atorvastatin to Reduce Inflammation in Acute Coronary Syndrome
Brief Title: COLchicine On-admission to Reduce Inflammation in Acute Coronary Syndrome (COLOR-ACS)
Acronym: COLOR-ACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda USL Toscana Centro (Other)
Responsible Party: Principal Investigator, Anna Toso, Cardiologist at the Santo Stefano Hospital, Prato, Italy, Azienda USL Toscana Centro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 20426; 2021-000637-13 (EudraCT Number)
Record Dates: First submitted 2022-02-08; First posted 2022-02-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: Colchicine; Atorvastatin; Acute Coronary Syndrome; C reactive protein; Acute Kidney Injury
MeSH Terms: conditions — Acute Coronary Syndrome; Acute Kidney Injury | interventions — Colchicine; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Participants are assigned to Colchicine plus standard treatment with Atorvastatin or only standard treatment with Atorvastatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine and Atorvastatin (Experimental): Colchicine 1 mg (0.5 mg for patients ≤ 70 Kg) on-admission followed by 0.5 mg/day until discharge plus Atorvastatin 80 mg on admission followed by 80 mg/day until discharge.
  Interventions: Drug: Colchicine; Drug: Atorvastatin
- Atorvastatin (Active Comparator): Atorvastatin 80 mg on admission followed by 80 mg/day until discharge.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Colchicine — Colchicine 1 mg (0.5 mg for patients ≤ 70 Kg) on-admission followed by 0.5 mg/day until discharge.
  Arms: Colchicine and Atorvastatin
Drug: Atorvastatin — Atorvastatin 80 mg on admission followed by 80 mg/day until discharge.

SUMMARY:
Since colchicine is known to have anti-inflammatory effects and inflammation is an early component of acute coronary syndrome (ACS), this study aims to evaluate the acute effects of low-dose colchicine, in addition to atorvastatin, administered on-admission to statin-naive patients with non-ST elevation ACS scheduled for early invasive strategy.

DETAILED DESCRIPTION:
On-admission all statin naive NSTEACS patients are randomized to receive either standard treatment of atorvastatin 80 mg or standard treatment plus colchicine (1 mg loading dose followed by 0.5 mg/day).

Inflammatory biomarker high sensitivity C reactive protein (hs-CRP) is measured in all patients on-admission and every 24 hours thereafter until discharge.

Cardiac and renal function parameters are evaluated to evidence the possible beneficial effects of the administration of colchicine in addition to atorvastatin alone both short- and medium-term (up to 30 days).

Colchicine tolerance is also investigated through monitoring for clinical side effects.

ELIGIBILITY:
Inclusion Criteria:

* non-ST elevation acute coronary syndrome;
* ≥ 18 years;
* statin-naive.

Exclusion Criteria:

* prior statin therapy and/or colchicine treatment;
* known allergy or hypersensitivity to colchicine or statins;
* current treatment with potent inhibitors of CYP3A4 or P-glycoprotein (eg., Cyclosporin, antiretroviral drugs, antimycotics, erythromicin and clarythromycin);
* previous or scheduled administration of any immunosuppressive therapy;
* known active malignancy;
* severe kidney disease (creatinine > 3 mg/dl or dialysis)
* severe liver disease (ALT and/or AST, > double ref. normal values in case of (a) total bilirubin > double ref. normal values, or (b) alteration in coagulation (INR> 1,5);
* severe heart failure (NYHA class ≥ 3 or cardiogenic shock) at hospital presentation;
* severe acute or chronic gastro-intestinal disease (nausea, vomiting, diarrhea, malabsorption disease, malnutrition);
* pregnancy or lactation;
* current COVID-19 or other infectious disease;
* refusal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
hsCRP change between admission and discharge | Average 4 days: from admission to discharge
  Effect of colchicine plus atorvastatin in limiting hsCRP changes compared to atorvastatin alone

SECONDARY OUTCOMES:
Delta variation in creatinine value from baseline to peak | Creatinine value is measured daily during hospitalization - average 4 days
  Delta variation (absolute and relative) in creatinine value from baseline value to peak value
Acute kidney injury incidence | Creatinine value is measured daily during hospitalization - average 4 days
  Creatinine increase >= 0.3 mg/dl within 48 hours after angiography
CK-MB peak value | CK-MB value is measured daily during hospitalization - average 4 days
  Comparison of CK-MB peak values in the two arms
Glomerular filtration rate changes at 30 days after discharge | Approximately 30 days
  Delta variation in the glomerular filtration rate from baseline to 30 days after discharge
Adverse clinical events from admission to 30 days after discharge | Approximately 30 days
  Myocardial infarction, glomerular filtration rate deterioration or all-cause death from admission to 30 days after discharge
Tolerance to colchicine | From admission to discharge - Approximately 4 days
  Percentage of patients who do not manifest side effects to colchicine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anna Toso, MD, Principal Investigator — Santo Stefano Hospital, Prato, Italy
Locations (3):
- Italy (3):
  - Gaia Chiara Selvaggia Magnaghi, Pescia
  - Marco Comeglio, Pistoia
  - Anna Toso, Prato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toso A, Leoncini M, Magnaghi G, Biagini F, Martini O, Maioli M, Villani S, Comeglio M, Bellandi F. Rationale and design of COLchicine On-admission to Reduce inflammation in Acute Coronary Syndrome (COLOR-ACS) study. J Cardiovasc Med (Hagerstown). 2023 Jan 1;24(1):52-58. doi: 10.2459/JCM.0000000000001389. Epub 2022 Nov 29. PMID 36473121